CLINICAL TRIAL: NCT04063397
Title: Persistent Postpartum Cardiovascular Dysfunction in Patients With Preeclampsia
Acronym: ECHO
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: Roche Diagnostics GmbH (Industry)
Responsible Party: Principal Investigator, Kara M Rood, MD, Assistant Professor, Maternal-Fetal Medicine, Ohio State University
Other Study IDs: 2018H0312
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Preeclampsia Severe or Mild; Cardiac Complication
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Echocardiography; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preeclampsia: 40 patients diagnosed with preeclampsia with or without severe features
  Interventions: Diagnostic Test: Echocardiogram; Diagnostic Test: Blood draw
- Control: 20 Control group of patients without hypertensive disorders of pregnancy
  Interventions: Diagnostic Test: Echocardiogram; Diagnostic Test: Blood draw

INTERVENTIONS:
Diagnostic Test: Echocardiogram — Serial echocardiograms will be done on all patients pre-delivery, and at 3-6 months
Diagnostic Test: Blood draw — Serial blood draws at same time points as echocardiograms for biomarker levels

SUMMARY:
The investigators plan to enroll women with PE prospectively to evaluate incremental cardiovascular risk in those who have PE with severe features. This study includes detailed echocardiographic evaluation at several time points. With the current proposal, the investigators aim to collect blood to evaluate several biomarkers to determine if there is a correlation with short and medium-term cardiovascular risk. This opens the door to earlier detection, treatment and improved cardiovascular outcomes.

DETAILED DESCRIPTION:
Preeclampsia (PE) is a multi-system progressive disorder affecting up to 8% of pregnancies. Epidemiologic studies have shown a significant association between PE and future cardiovascular disease (CVD) in women. Despite recognition of this relationship, there are no good markers to help determine which women are at highest risk, in particular as this relates to long-term cardiovascular risk, the number one cause of mortality in U.S. born women. As such, the study of PE and cardiovascular outcomes, in particular to identify early markers for the development of late CVD, provide insight into critical opportunities for early treatment and modification of disease trajectory in women.

The investigators plan to enroll women with PE prospectively to evaluate incremental cardiovascular risk in those who have PE with severe features. This study includes detailed echocardiographic evaluation at several time points. With the current proposal, the investigators aim to collect blood to evaluate several biomarkers to determine if there is a correlation with short and medium-term cardiovascular risk. This opens the door to earlier detection, treatment and improved cardiovascular outcomes.

The investigators hypothesize that preeclampsia with severe features confers a much higher risk of cardiovascular impairment compared to milder form of preeclampsia and healthy controls. If the hypothesis proves correct, these findings may change clinical practice by warranting routine echocardiogram for these patients for early recognition, intervention and treatment of cardiac dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Females older than 18 years of age
* Singleton pregnancy
* The patient is physically and mentally able to understand the informed consent and is willing to participate in this study
* Able to speak English
* Must meet one of the population categories, until each group has reached 20 subjects

Exclusion Criteria:

* Multiple gestation
* History of chronic hypertension or cardiac disease including but not limited to history of heart arrhythmias, congenital heart disease, and use of any cardiac medication (such as beta blockers, ACE inhibitors, calcium channel blockers) prior to pregnancy.
* History of medical problems that may contribute to cardiac dysfunction, including but not limited to chronic hypertension, poorly controlled hyperthyroidism and diabetes mellitus.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 40 patients with preeclampsia with or without severe features 20 control group patients with no hypertensive disorder of pregnancy
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Cardiac dysfunction | From delivery up to 3-6 months postpartum
  The following parameters will be measured to assess cardiac dysfunction:
  1. LV Size/function
     1. Biplane Method of Disks LVEF (a4C and 2C views for EDV and ESV)
     2. LV Fractional shortening- Septal thickness and PW thickness
     3. LV Strain- Basal longitudinal, Mid LV longitudinal, Apical LV longitudinal and Global LV longitudinal strain
     4. 3D LV EF
     5. Tei index
     6. Analysis of LV diastolic function- Mitral E wave, Mitral A wave, Mitral e', Mitral E/e', Mitral E/A and Mitral Decel time
  2. LA volume
  3. RA volume
  4. IVC size/compressibility with inspiration
  5. RV size/function
     1. RV length
     2. RV basal width
     3. RV FAC %
     4. TAPSE
     5. S'
     6. Tei index
     7. TR velocity
     8. RVSP
     9. TAPSE
     10. Longitudinal strain- Basal Longi, Basal longitudinal, Mid LV longitudinal, Apical LV longitudinal and Global LV longitudinal strain
  6. Basic valve assessment

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided